CLINICAL TRIAL: NCT00542932
Title: The Effects of a Home Exercise Video Programme for Patients With Chronic Obstructive Pulmonary Disease:Pilot Study
Brief Title: The Effects of a Home Exercise Video Programme for Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: University of Brighton (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/Q0703/151
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Exercise; Home
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (No Intervention)
- II (Active Comparator): Exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Watched Film A (promotional film)
  Film B (30 min exercise video) asked to to perform 4 times a week for 6 weeks at home
  Arms: II

SUMMARY:
Patients with COPD, suffer symptoms of breathlessness and leg weakness. Exercise programmes in the form of pulmonary rehabilitation (PR) have been shown to improve both of these symptoms significantly. PR involves patients attending a hospital or community centre. For some patients, leaving the house is an ordeal. This study investigated the effectiveness of an exercise video programme delivered in the patients home.

DETAILED DESCRIPTION:
Pulmonary Rehabilitation (PR) has been shown to deliver cost-effective improvements in dyspnoea, exercise tolerance and health-related quality of life (HRQoL) in people with chronic obstructive pulmonary disease (COPD). PR programmes in the United Kingdom (UK) are typically delivered on an outpatient basis, either at a hospital or suitable site in the community. It is not always possible however, for patients to access outpatient programmes due to lack of local availability or adequate transport from isolated locations. Severe breathlessness may reduce activity levels to such a degree that for many leaving the house is an ordeal. A British Lung Foundation (BLF) survey reported that less than 2% of UK COPD patients had access to a rehabilitation exercise programme, despite National Institute for Health and Clinical Excellence (NICE) and British Thoracic Society (BTS) recommendations that PR be made available to all patients who are functionally limited by dyspnoea. Meeting the demand for PR remains a challenge.

Access to the benefits of PR may be broadened if effective exercise could be administered at home. Current evidence suggests that home-based rehabilitation interventions result in smaller benefits as judged by exercise tolerance and quality of life when compared to supervised programmes. The impact of home based rehabilitation may be limited by multiple factors including, lack of health care professional supervision and lack of support from fellow COPD sufferers. This lack of support may lead to poor adherence to prescribed exercise intensity and frequency in home programmes.

One-to-one supervision on an individual basis is unlikely to be feasible or cost-effective, however, use of a home exercise video could enhance adherence to prescribed exercise programmes. Video media can be an effective means of delivering exercise instruction. No published research to date has investigated the effectiveness of a home exercise video for patients with COPD. We hypothesised that an exercise programme based on video instruction at home, could improve walking ability, breathlessness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Moderate/severe COPD
* Access to a video or DVD player

Exclusion Criteria:

* Comorbid condition that precludes safe exercise
* Previous attendance at a pulmonary rehabilitation programme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test | Baseline and 6 weeks

SECONDARY OUTCOMES:
Chronic Respiratory Disease Questionnaire | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Moxham, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom